CLINICAL TRIAL: NCT00728806
Title: Biomarker for Early Detection and Intervention of Peritoneal Ultrafiltration Failure
Brief Title: Biomarker for Peritoneal Ultrafiltration Failure
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Other Study IDs: SYSU-PROPDBM
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Continuous Ambulatory Peritoneal Dialysis
Keywords: Continuous Ambulatory Peritoneal Dialysis; Ultrafiltration failure; Biomarker; Proteomics

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples Without DNA — peritoneal tissue will be collected at the time of peritoneal dialysis catheter insertion or extubation. Serum and dialysate samples will be collected for protein analysis.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will examine the peritoneal tissue, serum and dialysate proteins of peritoneal dialysis (PD) patients with different types of peritoneal solute transport by differential proteomics techniques.

This study will be performed to identify the molecular difference between different types of peritoneal solute transport and explore biomarker for early detection as well as early intervention of peritoneal ultrafiltration failure.

DETAILED DESCRIPTION:
Ultrafiltration failure (UFF) is an important cause of technical failure in PD patients. It may develop over time and is, therefore, especially important in longterm PD. However, the study on UFF is very limited so far, there are still lack of biomarker for early detection and intervention of UFF.

Proteomics uses a rapidly evolving group of technologies to identify, quantify, and characterize a global set of proteins. It is characterized by high-throughput, high specificity and high-sensitivity. Therefore, proteomics has become a major focus of recent medical research.

This study will examine the peritoneal tissue, serum and dialysate proteins of continuous ambulatory peritoneal dialysis (CAPD) patients with different types of peritoneal solute transport by differential proteomics techniques. Correlation analysis will be used for the relationship between clinical data and the differential proteins, as well as verification of the differential proteins in the peritoneal tissue, serum and dialysate of patients with UFF. This study will be performed to identify the molecular difference between different types of peritoneal solute transport and explore biomarker for early detection as well as early intervention of peritoneal ultrafiltration failure.

ELIGIBILITY:
Inclusion Criteria:

* Continuous ambulatory peritoneal dialysis patients whose primary disease is chronic glomerulonephritis, The range of age is 20 to 65 year old.
* serum albumin level ≥ 35 g/L.
* Residual GFR ≥ 2 ml/min/1.73 m2.
* 500 ml/d ≤ urine output ≤ 1000 ml/d.
* Subjects who agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* Patients who are secondary nephropathy.
* Patients with congestive heart failure, angina, myocardial infarction, severe valvular heart disease, malignant hypertension, hypertensive encephalopathy or cerebrovascular accident.
* Patients with chronic liver disease, dyscrasia, psychiatric disorder, alcohol or drug abuse.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients and outpatients in the peritoneal dialysis center of 1st Affiliated Hospital, Sun Yat-Sen University
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, M.D. & Ph.D., Principal Investigator — 1st Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The 1st Affiliated Hospital, Sun Yet-sen University, Guangzhou, Guangdong, China